CLINICAL TRIAL: NCT03524950
Title: Effect of Dexmedetomidine on Stress Study of Pituitrin in Laparoscopic Hysteromyoma Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Xia CAO, student, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: D to stress study of pituitrin
Record Dates: First submitted 2018-05-02; First posted 2018-05-15 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Hysteromyoma
Keywords: stress; dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- no dexmedetomidine (No Intervention)
- high dose dexmedetomidine (Experimental)
  Interventions: Drug: Dexmedetomidine
- low dose dexmedetomidine (Experimental)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Ninety patients will be assigned to three groups. Group A add saline in general anesthesia laparoscopic hysteromyoma surgery. Group B add dexmedetomidine 1μg/Kg10minutes as loading dose, followed by 0.7μg/Kg/h for maintenance.Group C add dexmedetomidine 0.7μg/Kg10minutes as loading dose, followed by 0.5μg/Kg/h for maintenance.
  Arms: high dose dexmedetomidine; low dose dexmedetomidine

SUMMARY:
This study is about the effect of dexmedetomidine to the stress of pituitrin in laparoscopic hysteromyoma surgery. It is well known that pituitrin has been widespread used in the laparoscopic hysteromyoma surgery. Pituitrin includes oxytocin and vasopressin. Vasopressin increase body stress reaction through hypothalamic pituitary adrenal(HPA) axis. The HPA axis has has main role to the body stress reaction. Dexmedetomidine can inhibit the stress responses mediated by the sympathetic nervous system. Therefore,the effect of dexmedetomidine to the stress of pituitrin in laparoscopic hysteromyoma surgery is worth to be studied.

ELIGIBILITY:
Inclusion Criteria:

Surgery will be scheduled as first case in the morning at 9 Am. On arrival to the operation room, intravenous access will be achieved with venous cannula under local anesthesia with 2% lidocaine. Monitoring consisted of 5 lead electrocardiography, pulse oximeter, noninvasive blood pressure, end tidal carbon dioxide, and bispectral index.

Exclusion Criteria:

Diabetic,chronic hypertension,patients on drugs such as beta blockers or calcium channel blockers,pregnant or lactating women, patients with abnormal serum creatinine and blood urea nitrogen, and patients with a history of allergy to drugs particularly α2 agonists.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
acth | the acth before using pituitrin 5 minutes
  adrenocorticotropic hormone
acth | the acth after using pituitrin 20 minutes
  adrenocorticotropic hormone
acth | the acth after using pituitrin 120 minutes
  adrenocorticotropic hormone